CLINICAL TRIAL: NCT06722508
Title: Exercise and Nutritional Prehabilitation for Head and Neck Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2072911
Record Dates: First submitted 2024-11-19; First posted 2024-12-09 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Head Cancer; Neck Cancer; Sarcopenia; Head and Neck Cancer
Keywords: Exercise; Nutritional; Prehabilitation; Head; Neck; Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Sarcopenia; Motor Activity; Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- behavioral intervention (Experimental): The study involves a behavioral intervention (exercise and nutritional prehabilitation) designed to assess outcomes related to feasibility, acceptability, and safety in head and neck cancer patients. Outcomes are being measured following the intervention over a defined period (from diagnosis through 1-month post-surgery).
  Interventions: Behavioral: exercise and nutritional prehabilitation

INTERVENTIONS:
Behavioral: exercise and nutritional prehabilitation — The study involves a behavioral intervention (exercise and nutritional prehabilitation) designed to assess outcomes related to feasibility, acceptability, and safety in head and neck cancer patients. Outcomes are being measured following the intervention over a defined period (from diagnosis through 1-month post-surgery).

SUMMARY:
This study examines the acceptability, feasibility, and safety in developing a prehabilitation program for head and neck cancer patients. The purpose of this research is to access the safety and acceptability of using a prehabilitation program before head and neck cancer surgery.

DETAILED DESCRIPTION:
The purpose of this research is to access the safety and acceptability of using a prehabilitation program before head and neck cancer surgery. In this unblinded prospective study we will establish a 2-week prehabilitation program and assess whether this is feasible, acceptable to our patients, and safe. Subjects will be enrolled through August 2025, with a goal of enrolling 20 total subjects. The anticipated duration of each subject's involvement will be approximately 3 months, beginning at the time of their initial consultation and ending approximately 1 month after surgery.

Subjects will sign the informed consent form at initial visit and then receive a 2-week home- based exercise program to follow for the two weeks leading up to their surgical date. This exercise program will be provided both electronically through a link to our study-specific Med Bridge Program. Additionally, a hard-copy/PDF will be provided to the patients who prefer this format. Nutritional goals will be suggested, mainly with protein macronutrient goals defined as at least 1.2-2g/kg of protein per day.

At initial visit and the 1-month post-op visit, Timed Up and Go (TUG) and 6 Minute walk Test (6MWT) will be evaluated.

Subjects will begin the exercise program exactly two weeks (14 days) prior to surgery and will be instructed on their "start date" as soon as a surgical date is secured. Subjects will receive all necessary equipment (pedometer, resistance bands) from the study team, as well as a log-book for recording their compliance. The PI or designated study team-member will confirm with the subject this start-date, and perform weekly follow-up calls on day 7 and day 14 to monitor for any adverse events and compliance. Any report of increased pain related to the exercise program or injury will result in immediate recommendation for medical assessment and withdrawal from the study.

Standard-of-care cancer care will otherwise take place during the prehabilitation period, including any necessary laboratory and imaging testing. No additional testing will be required of the patient. Typically, patients are seen in an initial consultation and if surgery is recommended, preoperative labs and imaging are ordered if clinically necessary. Surgery date is typically within 3-4 weeks of initial consultation. If patients screen positive for malnutrition on the Malnutrition Screening Tool, standard-of-care referral to a dietician will be recommended.

Subjects will otherwise also have their usual post-operative and post-discharge care with their provider and have their final study-related visit approximately 1 month after surgery.

Primary end-point will be to assess the feasibility, acceptability, and safety of this program.2,3

- Safety will be monitored throughout the study period, including during the prehabilitation period with a study member calling the patient weekly (Day 7 and Day 14 or prehabilitation).

ELIGIBILITY:
Inclusion Criteria:

New head and neck cancer diagnosis Age > 18

Exclusion Criteria:

1. Prior treatment for head and neck cancer (surgery and/or radiation)
2. Acute or unstable cardiac conditions (unstable angina or symptomatic severe aortic stenosis)
3. American Society of Anesthesiologists physical status of 4 and 5
4. Disabling orthopedic or neuromuscular disease
5. Cardiac failure (New York Heart Association functional classes III and IV)
6. Severe chronic obstructive pulmonary disease
7. End-stage liver or kidney disease
8. Inability to swallow and/or feeding tube dependence
9. Any other comorbid medical, physical, and/or mental condition that contraindicates exercise or oral nutrition
10. Adults unable to consent
11. Age 17.99 or younger
12. Prisoners, pregnant women, or other vulnerable population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Completion Rate of 2-Week Prehabilitation Program | 2 weeks
  Percentage of participants who successfully complete the 2-week prehabilitation program for head and neck cancer patients.
Participant Safety During the 2-Week Program | 2 weeks
  Number of participants who experience adverse events during the 2-week prehabilitation program, assessed using CTCAE v5.0 criteria.
Acceptability of the Program | 2 weeks
  Number of participants who rate the prehabilitation program as acceptable, using a 5-point Likert scale (1 = Not Acceptable, 5 = Very Acceptable).
Feasibility of the Program | 2 weeks
  Percentage of planned exercise and nutrition activities completed by participants during the 2-week prehabilitation program.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne S Abouyared, MD, Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - UC Davis Health, Sacramento, California
  - UC Davis Medical Center, Sacramento, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Powell R, Davies A, Rowlinson-Groves K, French DP, Moore J, Merchant Z. Acceptability of prehabilitation for cancer surgery: a multi-perspective qualitative investigation of patient and 'clinician' experiences. BMC Cancer. 2023 Aug 11;23(1):744. doi: 10.1186/s12885-023-10986-0. PMID 37568097
- [Background] Knols R, Aaronson NK, Uebelhart D, Fransen J, Aufdemkampe G. Physical exercise in cancer patients during and after medical treatment: a systematic review of randomized and controlled clinical trials. J Clin Oncol. 2005 Jun 1;23(16):3830-42. doi: 10.1200/JCO.2005.02.148. PMID 15923576

DOCUMENTS (1):
  • Informed Consent Form (2023-11-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT06722508/ICF_000.pdf